CLINICAL TRIAL: NCT06975202
Title: Test-retest Reliability and Agreement of Trunk Muscle Activation in Pain-free Persons
Acronym: MAS-Reliab
Status: Recruiting | Type: Observational
Sponsor: University Ghent (Other)
Collaborators: VZW Educatieve Lichaamsbeweging (Unknown)
Responsible Party: Sponsor
Other Study IDs: B6702022000426
Record Dates: First submitted 2024-09-20; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Controls; Healthy Control
Keywords: reliability; agreement; muscle activation; functional tasks

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pain-free persons: Pain-free persons
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The aim of the study is to investigate test-retest reliability and agreement of trunk muscle activation during functional tasks and clinical sensorimotor control tests in pain-free persons.

DETAILED DESCRIPTION:
Optimal muscle function is essential for daily life functioning. The current literature suggests that alterations in trunk muscle activation might be one of the contributing factors to the persistence and recurrence of musculoskeletal disorders, including low back pain and lower limb injuries. It is crucial that trunk muscle activation during functional tasks has sufficient reliability and agreement to interpret (longitudinal) studies.

A limited number of studies have investigated the reliability and agreement of trunk muscle activation during dynamic (functional) tasks. Moreover, all these studies used simple discrete outcomes such as mean or peak amplitude. An important limitation is that these single zero-dimensional outcome values ignore the temporal aspects of dynamic tasks. As such, potentially relevant time-specific characteristics of muscle activation might be missed. A comprehensive reliability analysis of curve data (i.e., one-dimensional data) that considers the temporal timeframe is therefore required. An overview of reliability analyses of curve data can be found in Pini et al. This paper concluded that integrated pointwise indices can be recommended. Recently, this innovative analysis was used in biomechanical studies investigating the kinematics and kinetics during jump landing. However, to the best of our knowledge, integrated pointwise indices have not been used to determine reliability and agreement of muscle activation during functional tasks.

The lumbar multifidus has received extensive attention over the past 25 years. The multifidus muscle consists of deep and short fibers that overlay up to 2 segments (i.e., deep multifidus) and more superficial and longer fibers that cross up to 5 segments (i.e., superficial multifidus). As a result of their anatomy, the deep multifidus (DM) predominantly provides segmental stabilization through compressive forces, while the superficial multifidus (SM) mainly generate lumbar movement (i.e., extension, lateral bending, and rotation). Previous studies showed that the distinction between DM and SM activation is especially important for persons with low back pain. Although the results in persons with low back pain vary, the current literature shows a trend towards an overall reduced activation of the DM, while the activation of the SM is often augmented. As such, a clinical test that assesses voluntary DM activation has been proposed and specific motor control therapy that targets the DM has been shown to reduce pain and disability in patients with low back pain. Fine-wire electromyography (EMG) is the only technique that is able to record selective deep muscle activation during dynamic functional tasks, as opposed to other techniques such as surface EMG. However, reliability studies that use fine-wire EMG to measure selective DM and SM activation during functional tasks are currently lacking.

Therefore, this study aims to investigate test-retest reliability and agreement of trunk muscle activation measured with surface and fine-wire EMG during functional tasks in pain-free persons.

ELIGIBILITY:
Inclusion Criteria:

- Pain-free persons between 18 and 65 years old

Exclusion Criteria:

* Persons experiencing low back pain in the past year
* Patients with serious underlying conditions (e.g., multiple sclerosis)
* Previous spinal surgery
* Persons with any type of blood clotting disorder
* Persons with upper-limb complaints that prevent them from exerting (maximum) force with their arms or hands.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pain-free persons will be recruited through online advertisement, flyers and posters.
Sampling Method: Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Trunk muscle onset during the rapid arm movement test | Baseline (test-session)
  Trunk muscle onset latencies in response to the unilateral rapid arm movement test will be measured by means of electromyography.
Trunk muscle onset during the rapid arm movement test | After a 30-minute break (retest-session)
  Trunk muscle onset latencies in response to the unilateral rapid arm movement test will be measured by means of electromyography.

SECONDARY OUTCOMES:
Trunk muscle (co-)activation | Baseline (test-session)
  The participant sits on a stool and holds a horizontal bar with both hands, shoulders at 90 degrees (arms are horizontal). The horizontal bar is secured to the ground using a rope and weights. The participant pushes the horizontal bar upwards without moving the arms, pelvis, or spine. The activation of the back and abdominal muscles will be further investigated.
Trunk muscle (co-)activation | After a 30-minute break (retest-session)
  The participant sits on a stool and holds a horizontal bar with both hands, shoulders at 90 degrees (arms are horizontal). The horizontal bar is secured to the ground using a rope and weights. The participant pushes the horizontal bar upwards without moving the arms, pelvis, or spine. The activation of the back and abdominal muscles will be further investigated.
Back muscle activation | Baseline (test-session)
  Back muscle activation will be analyzed during (1) bilateral reaching in standing position, (2) unilateral/bilateral reaching starting in neutral sitting position, and (3) unilateral/bilateral reaching starting in habitual sitting position.
Back muscle activation | After a 30-minute break (retest-session)
  Back muscle activation will be analyzed during (1) bilateral reaching in standing position, (2) unilateral/bilateral reaching starting in neutral sitting position, and (3) unilateral/bilateral reaching starting in habitual sitting position.
Voluntary multifidus activation | Baseline (test-session)
  Voluntary multifidus activation will be measured while the participant lies prone on a treatment table. The participant will be instructed to gently activate the multifidus muscle without movement of the pelvis or spine, while breathing is maintained.
Voluntary multifidus activation | After a 30-minute break (retest-session)
  Voluntary multifidus activation will be measured while the participant lies prone on a treatment table. The participant will be instructed to gently activate the multifidus muscle without movement of the pelvis or spine, while breathing is maintained.
Involuntary multifidus activation | Baseline (test-session)
  Involuntary multifidus activation will be assessed by means of the multifidus lift test (Hebert et al., 2015). The participant is lying in the prone position with the shoulders in 120° abduction and 90° flexion at the elbows. The participant will be asked to lift the entire arm approximately 5 cm from the treatment table. The multifidus activation on the contralateral side will be investigated further.
Involuntary multifidus activation | After a 30-minute break (retest-session)
  Involuntary multifidus activation will be assessed by means of the multifidus lift test (Hebert et al., 2015). The participant is lying in the prone position with the shoulders in 120° abduction and 90° flexion at the elbows. The participant will be asked to lift the entire arm approximately 5 cm from the treatment table. The multifidus activation on the contralateral side will be investigated further.

CONTACTS AND LOCATIONS:
Overall Officials: Lieven Danneels, Professor, Principal Investigator — University Ghent
Locations (1):
- Faculty of Medicine and Health Sciences, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Moseley GL, Hodges PW, Gandevia SC. External perturbation of the trunk in standing humans differentially activates components of the medial back muscles. J Physiol. 2003 Mar 1;547(Pt 2):581-7. doi: 10.1113/jphysiol.2002.024950. Epub 2002 Dec 20. PMID 12562944
- [Background] MacDonald D, Moseley GL, Hodges PW. People with recurrent low back pain respond differently to trunk loading despite remission from symptoms. Spine (Phila Pa 1976). 2010 Apr 1;35(7):818-24. doi: 10.1097/BRS.0b013e3181bc98f1. PMID 20228708
- [Background] Schelin L, Pini A, Markstrom JL, Hager CK. Test-retest reliability of entire time-series data from hip, knee and ankle kinematics and kinetics during one-leg hops for distance: Analyses using integrated pointwise indices. J Biomech. 2021 Jul 19;124:110546. doi: 10.1016/j.jbiomech.2021.110546. Epub 2021 Jun 12. PMID 34171677
- [Background] Pini A, Markstrom JL, Schelin L. Test-retest reliability measures for curve data: an overview with recommendations and supplementary code. Sports Biomech. 2022 Feb;21(2):179-200. doi: 10.1080/14763141.2019.1655089. Epub 2019 Oct 3. PMID 31578129
- [Background] Wildenbeest MH, Kiers H, Tuijt M, van Dieen JH. Reliability of measures to characterize lumbar movement patterns, in repeated seated reaching, in a mixed group of participants with and without low-back pain: A test-retest, within- and between session. J Biomech. 2021 May 24;121:110435. doi: 10.1016/j.jbiomech.2021.110435. Epub 2021 Apr 15. PMID 33894470
- [Background] Matheve T, Hodges P, Danneels L. The Role of Back Muscle Dysfunctions in Chronic Low Back Pain: State-of-the-Art and Clinical Implications. J Clin Med. 2023 Aug 24;12(17):5510. doi: 10.3390/jcm12175510. PMID 37685576
- [Background] Hodges PW, Danneels L. Changes in Structure and Function of the Back Muscles in Low Back Pain: Different Time Points, Observations, and Mechanisms. J Orthop Sports Phys Ther. 2019 Jun;49(6):464-476. doi: 10.2519/jospt.2019.8827. PMID 31151377
- [Background] Hebert JJ, Koppenhaver SL, Teyhen DS, Walker BF, Fritz JM. The evaluation of lumbar multifidus muscle function via palpation: reliability and validity of a new clinical test. Spine J. 2015 Jun 1;15(6):1196-202. doi: 10.1016/j.spinee.2013.08.056. Epub 2013 Oct 4. PMID 24314767